CLINICAL TRIAL: NCT06643728
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study of Bimagrumab and Tirzepatide, Alone or in Combination, to Investigate the Efficacy and Safety in Adult Participants With Obesity or Overweight Without Type 2 Diabetes
Brief Title: A Study to Investigate Weight Management With Bimagrumab (LY3985863) and Tirzepatide (LY3298176), Alone or in Combination, in Adults With Obesity or Overweight
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27265; J4Z-MC-GIDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight
Keywords: Muscle; Lean; Fat
MeSH Terms: conditions — Obesity; Overweight; Platelet Glycoprotein IV Deficiency | interventions — bimagrumab; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A: Bimagrumab Dose 2 + Tirzepatide Placebo (Experimental): Participants will receive bimagrumab subcutaneously (SC) and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide Placebo
- Part A: Bimagrumab Placebo + Tirzepatide Dose 1 (Active Comparator): Participants will receive bimagrumab placebo SC and tirzepatide SC
  Interventions: Drug: Tirzepatide; Drug: Bimagrumab Placebo
- Part A: Bimagrumab Placebo + Tirzepatide Dose 2 (Active Comparator): Participants will receive bimagrumab placebo SC and tirzepatide SC
  Interventions: Drug: Tirzepatide; Drug: Bimagrumab Placebo
- Part A: Bimagrumab Dose 1 + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part A: Bimagrumab Dose 1 + Tirzepatide Dose 2 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part A: Bimagrumab Dose 2 + Tirzepatide Dose 2 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part A: Bimagrumab Placebo + Tirzepatide Placebo (Placebo Comparator): Participants will receive bimagrumab placebo SC and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab Placebo; Drug: Tirzepatide Placebo
- Part B: Bimagrumab Dose 2 (no titration) + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part B: Bimagrumab Dose 2 (fast titration) + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part B: Bimagrumab Dose 2 (slow titration) + Tirzepatide Dose 1 (Experimental): Participants will receive bimagrumab SC and tirzepatide SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide
- Part B: Bimagrumab Dose 1 + Tirzepatide Placebo (Experimental): Participants will receive bimagrumab SC and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab; Drug: Tirzepatide Placebo
- Part B: Bimagrumab Placebo + Tirzepatide Placebo (Placebo Comparator): Participants will receive bimagrumab placebo SC and tirzepatide placebo SC
  Interventions: Drug: Bimagrumab Placebo; Drug: Tirzepatide Placebo

INTERVENTIONS:
Drug: Bimagrumab — Administered SC
  Other Names: LY3985863; BYM338; VER201
  Arms: Part A: Bimagrumab Dose 1 + Tirzepatide Dose 1; Part A: Bimagrumab Dose 1 + Tirzepatide Dose 2; Part A: Bimagrumab Dose 2 + Tirzepatide Dose 2; Part A: Bimagrumab Dose 2 + Tirzepatide Placebo; Part B: Bimagrumab Dose 1 + Tirzepatide Placebo; Part B: Bimagrumab Dose 2 (fast titration) + Tirzepatide Dose 1; Part B: Bimagrumab Dose 2 (no titration) + Tirzepatide Dose 1; Part B: Bimagrumab Dose 2 (slow titration) + Tirzepatide Dose 1
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Part A: Bimagrumab Dose 1 + Tirzepatide Dose 1; Part A: Bimagrumab Dose 1 + Tirzepatide Dose 2; Part A: Bimagrumab Dose 2 + Tirzepatide Dose 2; Part A: Bimagrumab Placebo + Tirzepatide Dose 1; Part A: Bimagrumab Placebo + Tirzepatide Dose 2; Part B: Bimagrumab Dose 2 (fast titration) + Tirzepatide Dose 1; Part B: Bimagrumab Dose 2 (no titration) + Tirzepatide Dose 1; Part B: Bimagrumab Dose 2 (slow titration) + Tirzepatide Dose 1
Drug: Bimagrumab Placebo — Administered SC
  Arms: Part A: Bimagrumab Placebo + Tirzepatide Dose 1; Part A: Bimagrumab Placebo + Tirzepatide Dose 2; Part A: Bimagrumab Placebo + Tirzepatide Placebo; Part B: Bimagrumab Placebo + Tirzepatide Placebo
Drug: Tirzepatide Placebo — Administered SC
  Arms: Part A: Bimagrumab Dose 2 + Tirzepatide Placebo; Part A: Bimagrumab Placebo + Tirzepatide Placebo; Part B: Bimagrumab Dose 1 + Tirzepatide Placebo; Part B: Bimagrumab Placebo + Tirzepatide Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of Bimagrumab and Tirzepatide, alone or in combination, in adults with obesity or overweight, with at least one obesity related comorbidity, without Type 2 Diabetes. The study will last about 70 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of

  * ≥30 kilograms per square meter (kg/m2) or
  * ≥27 kg/m2 and <30 kg/m2, with at least one of the following weight-related comorbidities:

    * Hypertension
    * Dyslipidemia
    * Cardiovascular disease
    * Obstructive sleep apnea
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss)

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity
* Have at least one laboratory value suggestive of diabetes during screening
* Use of metformin, or any other glucose-lowering medications
* Have Type 1 Diabetes, latent autoimmune diabetes, been diagnosed with any form of diabetes mellitus except for a prior diagnosis of gestational diabetes mellitus, or history of ketoacidosis or hyperosmolar coma
* Have poorly controlled hypertension
* Have any of the following cardiovascular conditions within 3 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have ongoing or a history of frequent intermittent or chronic tachyarrhythmia syndromes
* Have ongoing or a history of bradyarrhythmias other than sinus bradycardia
* Have a history of New York Heart Association (NYHA) Functional Classification III or IV congestive heart failure
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have signs and symptoms of any liver disease
* Have a disease or condition known to cause gastrointestinal malabsorption or a known clinically significant gastric emptying abnormality
* Have a history of acute or chronic pancreatitis
* Have renal impairment, measured as estimated glomerular filtration rate <30 mL/minute/1.73 m2
* Currently taking or have taken medications that may cause significant weight gain or promote weight loss within 3 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 24

SECONDARY OUTCOMES:
Percent Change from Baseline in Total Body Fat Mass by Dual-Energy X-Ray Absorptiometry (DXA) | Baseline, Week 24, Week 48
Change from Baseline in Body Weight | Baseline, Week 24, Week 48
Percentage of Participants Achieving ≥5% Body Weight Reduction | Baseline, Week 24, Week 48
Percentage of Participants Achieving ≥10% Body Weight Reduction | Baseline, Week 24, Week 48
Percentage of Participants Achieving ≥15% Body Weight Reduction | Baseline, Week 24, Week 48
Change from Baseline in Waist Circumference | Baseline, Week 24, Week 48
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 24, Week 48
Change from Baseline in Waist-to-Height Ratio (WHtR) | Baseline, Week 24, Week 48
Percent Change from Baseline in Visceral Adipose Tissue (VAT) | Baseline, Week 24, Week 48
Percent Change from Baseline in Total Body Lean Mass by DXA | Baseline, Week 24, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Central Research Associates, Birmingham, Alabama
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Suncoast Research Group, Miami, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study to Investigate Weight Management With Bimagrumab (LY3985863) and Tirzepatide (LY3298176), Alone or in Combination, in Adults With Obesity or Overweight — https://trials.lilly.com/en-US/trial/546217